CLINICAL TRIAL: NCT06616337
Title: Retrospective Study of the Acceptability and Effectiveness of a Dialectical Behavioral Therapy Group in Patients Suffering From Emotional Dysregulation (Borderline Personality Disorder, Bipolar Disorder and Adult ADHD)
Brief Title: Patients Suffering From Emotional Dysregulation
Acronym: Dys-Emotion
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9137
Record Dates: First submitted 2024-05-21; First posted 2024-09-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-05

CONDITIONS: Emotional Dysregulation
Keywords: Emotional Dysregulation; Schizophrenia; Bipolar disorder; Borderline personality disorder; Attention deficit hyperactivity disorder (ADHD)
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Borderline Personality Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Emotional dysregulation (ED) is a common syndrome in psychiatric disorders. It is characterized by intense emotions, easily triggered, and with significant psychological impact: explosions of anger, irritability, impulsivity, emotional lability, etc. It is systematic in borderline personality disorder, and observed in a majority of patients with bipolar disorder. (even in the interictal period), adult ADHD, or addictions. ED is a cause of psychological distress, suicidal behavior or non-suicidal self-injury, and impaired quality of life. Pharmacological treatments only very partially improve these symptoms. Psychotherapies aimed at reducing ED are poorly developed in France. Dialectical behavioral therapy is a therapy that has shown its effectiveness in ED of BPD.

This is why the psychiatry and addiction center of the University Hospitals of Strasbourg has set up groups using this psychotherapeutic approach based on this technique for almost 3 years. This technique being very little practiced in France, and even less studied, we want to see if it is adapted to a French population not accustomed to this type of practice.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Having participated in the first session of a GREMO group, which is a behavioral and dialectical therapy protocol from January 1, 2018 to December 31, 2023,
* Subject not opposing the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Subject having expressed their opposition to the reuse of their personal data for scientific research purposes.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) having participated in the first session of a GREMO group, which is a behavioral and dialectical therapy protocol during the period from January 1, 2018 to December 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01-21 (Estimated)

PRIMARY OUTCOMES:
Evaluate the change of symptoms of emotional dysregulation | Up to 1 year
  * The assessment is based on the DERS scale. Participants are asked to indicate how often the items apply to themselves, with responses ranging from 1 to 5,
  * The score between :
    * 1 means almost never (0 to 10%),
    * 2 means sometimes (11 to 35%),
    * 3 means about half the time (36 to 65%),
    * 4 means most of the time (66 to 90%),
    * 5 means almost always (91 to 100%).

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Psychiatrie 2 - CHU de Strasbourg - France, Strasbourg, France